CLINICAL TRIAL: NCT00155103
Title: Effect of Polymorphisms in the IL-1 Gene Complex on the Development of Chronic Hepatitis and Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361700927; NSC 93-2314-B-002-226
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2005-07

CONDITIONS: Hepatitis B; Carcinoma, Hepatocellular; Polymorphism, Genetic
Keywords: Hepatitis B; Carcinoma, Hepatocellular; Polymorphism, Genetic
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine the effect of polymorphisms in the IL-1 gene complex on the development of chronic hepatitis and hepatocellular carcinoma.

DETAILED DESCRIPTION:
We analyzed single-nucleotide polymorphisms in the genes for interleukin-1a, interleukin-1b, interleukin-1-receptor antagonist, interleukin-1-receptor type I, and interleukin-1-receptor type II in 400 normal control and patients (chronic hepatitis and hepatocellular carcinoma). Genotypes were tested for an association with development of chronic hepatitis and hepatocellular carcinoma by multivariable analysis. A second cohort of 1200 normal control and patients (chronic hepatitis and hepatocellular carcinoma) was independently analyzed for the genotype associations identified in the first cohort.

ELIGIBILITY:
Inclusion Criteria:

* Normal controls
* Cases of chronic hepatitis and hepatocellular carcinoma

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Li-Hui Tseng, M.D., Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- Department of Medical Genetics; National Taiwan University Hospital, Taipei, Taipei, Taiwan